CLINICAL TRIAL: NCT03918824
Title: Retrospective Analysis of the Influence of Iodinated Contrast Volume Injected During Coronarography on Contrast Nephropathy.
Brief Title: Influence of Iodinated Contrast Volume Injected During Coronarography on Contrast Nephropathy.
Status: Completed | Type: Observational
Sponsor: Agnieszka Pozdzik (Other)
Responsible Party: Sponsor-Investigator, Agnieszka Pozdzik, Head of nephro-dialysis clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Bensliman
Record Dates: First submitted 2019-03-26; First posted 2019-04-18 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Nephropathy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
Coronary heart disease remains one of the main causes of death in the world. One of the treatments for coronary heart disease is percutaneous coronary intervention (PCI). This requires the arterial administration of iodinated contrast medium (ICP) to visualize the state of the coronary arteries and possibly apply the treatment.

For the vast majority of the population, exposure to ICP is perfectly well tolerated. Nevertheless, some complications can occur including a nephropathy induced by the injection of a contrast product (NIC). NIC is the third cause of an acquired acute renal failure within the hospital.It significantly increases morbidity and mortality and prolongs the hospital stay.

Of all the procedures requiring ICP administration, PCI is associated with the highest rate of NIC.This evidence is explained by the fact that patients benefiting from such exploration have a higher risk profile in terms of cardiovascular comorbidities and associated pathologies.Age, preexisting alteration of renal function, diabetes mellitus, polypharmacy, congestive heart failure, type and volume of iodinated contrast medium are the main risk factors for developing NIC.

Nowadays, the use of PCI in the assessment of coronary heart disease in patients with these risk factors is becoming more frequent. This is linked to the aging of the population and the increasing incidence of cardiovascular diseases.

ICP-induced nephrotoxicity results from two main phenomena: the renal medullary hypoxia caused by the vasoconstriction of peritubular capillaries and a direct cytotoxicity towards tubular epithelial cells.These intra-renal mechanisms lead to an acute renal function impairment.NIC is defined as an increase of serum creatinemia ≥ 0.5 mg / dL (or a 25% increase) from the baseline in the 48-72h following PC injection with no other obvious etiology. It reaches its peak between the 3rd and 5th day with a resolution in 10 to 21 days.

The prevention of NIC based primarily on the identification of patients at risk and the use of pharmacological means (as hydration protocol). In contrast, there is little data on the relationship between NIC and the PCI volume used. To the investigator's knowledge, the threshold of toxic volume is not well defined. Taking into account these elements, the investigators propose to study the relation between the volume of iodinated contrast product injected during an ICP and the occurrence of a NIC according to the criteria mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who have undergone percutaneous coronary intervention with contrast medium Xenetic (Lobitridol ®) in the CHU Brugmann Hospital coronary angiography unit since 2013
* Access to extensive demographic, clinical and biological data

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who have undergone percutaneous coronary intervention with contrast medium Xenetic (Lobitridol ®) in the CHU Brugmann Hospital coronary angiography unit since 2013.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
incidence of nephropathies induced by the injection of iodinate contrast medium | 7 years
  incidence of nephropathy induced by injection of contrast medium
Volume of iodinated contrast medium injected | 1 day
  Volume of iodinated contrast medium injected
Body mass | 1 day
  Body mass
Urea concentration | 10 days after PCI
  Urea concentration
Creatinin rate | 10 days after PCI
  Creatinin rate
Glomerular filtration rate | 10 days after PCI
  Glomerular filtration rate

SECONDARY OUTCOMES:
Existence of risk factors (yes/no) | 7 years
  Existence of at least one of these risk factors: diabetes mellitus, abnormal blood pressure, abnormal kidney function, congestive heart failure.
Urea concentration | Baseline (day of percutaneous coronary intervention (PCI))
  Urea concentration
Urea concentration | 24 hours after of PCI
  Urea concentration
Urea concentration | 48 hours after PCI
  Urea concentration
Urea concentration | 72 hours after PCI
  Urea concentration
Urea concentration | 21 days after PCI
  Urea concentration
Urea concentration | 1 year after PCI
  Urea concentration
Creatinin rate | Baseline (day of percutaneous coronary intervention (PCI))
  Creatinin rate
Creatinin rate | 24 hours after of PCI
  Creatinin rate
Creatinin rate | 48 hours after PCI
  Creatinin rate
Creatinin rate | 72 hours after PCI
  Creatinin rate
Creatinin rate | 21 days after PCI
  Creatinin rate
Creatinin rate | 1 year after PCI
  Creatinin rate
Glomerular filtration rate | Baseline (day of percutaneous coronary intervention (PCI))
  Glomerular filtration rate
Glomerular filtration rate | 24 hours after of PCI
  Glomerular filtration rate
Glomerular filtration rate | 48 hours after PCI
  Glomerular filtration rate
Glomerular filtration rate | 72 hours after PCI
  Glomerular filtration rate
Glomerular filtration rate | 21 days after PCI
  Glomerular filtration rate
Glomerular filtration rate | 1 year after PCI
  Glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bensliman, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No